CLINICAL TRIAL: NCT03624023
Title: A Pilot Phase I/II Study to Evaluate the Safety and Efficacy of TWB-103 in Treating Lower Limb Ulcers on Patients With Diabetes Mellitus
Brief Title: TWB-103 for Treating Lower Limb Ulcers on Patients With DM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Transwell Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-FDF-C002
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TWB-103 (Experimental): (Mixture of TWB-102 cell and TWB-103 hydrogel)
  Interventions: Drug: TWB-103

INTERVENTIONS:
Drug: TWB-103 — TWB-103 will be applied to the target ulcer wound once a week by the investigator, starting from Day 1, until wound closure is confirmed or up to 12 weekly applications
  Other Names: Mixture of TWB-102 cell and TWB-103 hydrogel

SUMMARY:
Primary Objective:

To assess the safety profile of TWB-103 administered to subjects with diabetic lower limb ulcers

Secondary Objective:

To explore the efficacy of TWB-103 administered to subjects with diabetic lower limb ulcers

DETAILED DESCRIPTION:
Diabetic foot ulcers are primarily caused by poor circulation, high blood sugar (hyperglycemia), nerve damage, and foot irritation or injury. These factors, particularly poor circulation and high blood sugar, often hinder the healing process of ulcers. TWB-103 is a combination of TWB-102 cells (human fetal dermal fibroblasts) and TWB-103 hydrogel. The objective of this study was to determine whether the application of TWB-103 on diabetic ulcer wounds could accelerate the healing process in subjects with diabetic lower limb ulcers that had not shown signs of healing for at least four weeks. The study was designed as a Phase I/II, single-arm trial, with a planned enrollment of 10 subjects. These subjects would receive up to 12 weekly applications of TWB-103, and the study would evaluate both the safety and efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 20 years of age.
2. With diagnosed diabetic mellitus (DM), e.g. currently under DM medication treatment, or with HbA1c ≧6.5% but < 12%, or with fasting plasma glucose ≧126 mg/dL (7.0 mmol/L), or with plasma glucose ≧ 200 mg/dL (11.1 mmol/L) in the two-hour 75-gram oral glucose tolerance test (OGTT).
3. With at least one cutaneous ulcer on the foot or the lower legs, and not healing for at least 4 weeks (the ≧2-week standard of care period can be counted as part of the 4-week ulcer history).
4. With ankle brachial index (ABI) ≥ 0.4 on the limb with the study ulcer. For subjects with 0.6>ABI ≧0.4, the investigator will arrange for providing proper treatment to the subject, such as improving circulation by medication or surgical procedures, etc.
5. The study wound is not prone to infection.
6. The wound should allow complete sealing of the wound by TegadermTM film.
7. The study wound size is between 1~33 cm2. The depth of wound may reach ligament, joint capsule, fascia, or tendon. There should be no sign of osteomyelitis. The wound does not exceed Wagner Grade 27.
8. Under the standard care of Investigator for at least 2 weeks, the study wound has not shown significant healing. Significant healing is defined as the following: The area of healed tissue reaches at least 30% of the area of initially presented wound.
9. When the subject has more than one wound which met the inclusion criteria, only one wound is selected as the study wound. The other wounds will be treated by standard cares.
10. Co-morbidities are under control and non-life threatening as determined by the Investigator based on medical history, physical examination, vital signs, or clinical laboratory tests, etc.
11. A negative pregnancy test at Screening. This applies to any female subject with childbearing potential.
12. Agrees to use acceptable contraceptive methods while on study (from signing informed consent form to the end of the study). This applies to any female subject with childbearing potential and any male subject whose female partner has childbearing potential.

    Acceptable contraceptive methods include:
    1. Established use of oral, injected or implanted hormonal methods of contraception
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps)
13. Able to follow the Investigator's instruction on wound care.
14. With signed informed consent form.

Exclusion Criteria:

1. Being pregnant or nursing.
2. With autoimmune disease other than diabetes, e.g. lupus erythematosus, multiple sclerosis.
3. With current malignancy or hypo-immunity.
4. With history of recurrent cancer, metastatic cancer, cancer which has high probability of metastasis, or cancer on the limb where the study wound is located.
5. With serum chemistry abnormalities below

   1. AST or ALT > 5 × ULN,
   2. Serum albumin < 2.0 g/dL,
6. With history of HIV infection
7. With history of alcoholism or drug abuse.
8. Received any cell-based product at the study wound.
9. Received an investigational drug, device or biological/bioactive treatment within 30 days prior to Screening Visit.
10. With any clinical condition or significant concurrent disease judged by the investigator to complicate the evaluation of the trial treatment.
11. With history of sensitivity to materials of bovine, porcine origin, or human serum albumin.
12. With active infection or active osteomyelitis in the study wound.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niann-Tzyy Dai, PhD, Principal Investigator — Tri-Service General Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed in a Phase I/II, single-arm manner. This study planned to enroll 10 subjects (including 8 evaluable per-protocol subjects) with diabetic lower limb ulcers for treating with up to 12 weekly applications of TWB-103 and evaluating the safety and efficacy.
Pre-assignment Details: Eligibility was checked during screening and at Day 1 Visit. The potential subjects with diabetic lower limb ulcer were arranged to receive standard of care only for at least 2 weeks during screening period. The standard of care was performed at the investigator's discretion based on the condition of each subject. Any subject whose study ulcer size decreases by 30% or more after this standard of care was excluded from the study.
Period: Overall Study
Arm/Group | TWB-103
Started | 10
Completed | 6
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Arm/Group | TWB-103
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (18.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 10
Sum of Target Ulcer Surface Area [Mean (Standard Deviation); unit: cm^2]
  Sum of Target Ulcer Surface Area before Standard-of-Care | 3.1 (2.42)
  Sum of Target Ulcer Surface Area after Standard-of-Care | 2.8 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Pre-existing abnormalities are considered as AE or SAE only when the conditions escalate. The following events should be discussed specifically:
  1. Study wound and its periphery: Infection, pain, pruritus/irritation, skin dysfunction/blister, osteomyelitis, cellulitis, edema/swelling and unexpected surgery.
  2. Non-study area and systemic: Infection, pain, pruritus/irritation, skin dysfunction/blister, osteomyelitis, cellulitis, edema/swelling, unexpected surgery, accidental injury, abnormal lab test and general disorders.
Time Frame: Day 1~ Day 169
Population: All Subject Population.
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103
Number analyzed (Participants) | 10
Participants
  AEs | 8
  SAEs | 3

2. Secondary Outcome: The Percentage of Subjects With Confirmed Study Wound Closure at Each Week up to 12 Weeks.
Description: Wound closure is defined as "full epithelialization of the wound with the absence of drainage and without sign of abscess under the epithelium". An ulcer is considered healed only after wound closure is re-confirmed at the visit 2 weeks later.
Time Frame: Week 1 ~ Week 12
Population: All Subject Population.
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103
Number analyzed (Participants) | 10
Participants
  Adjusted Visit 3 (Week 1) with LOCF | 0
  Adjusted Visit 4 (Week 2) with LOCF | 0
  Adjusted Visit 5 (Week 3) with LOCF | 1
  Adjusted Visit 6 (Week 4) with LOCF | 1
  Adjusted Visit 7 (Week 5) with LOCF | 1
  Adjusted Visit 8 (Week 6) with LOCF | 2
  Adjusted Visit 9 (Week 7) with LOCF | 2
  Adjusted Visit 10 (Week 8) with LOCF | 3
  Adjusted Visit 11 (Week 9) with LOCF | 5
  Adjusted Visit 12 (Week 10) with LOCF | 5
  Adjusted Visit 13 (Week 11) with LOCF | 6
  Adjusted Visit 14 (Week 12) with LOCF | 6

3. Secondary Outcome: Time to Confirmed Wound Closure for Those Subjects Whose Wounds Are Healed During Treatment Period and During the Study Period.
Description: as for outcome 2
Time Frame: Week 1 ~ Week 12
Population: All Subject Population.
  Median time to confirmed ulcer closure up to EOS (End of Study) was also 70 days (Range: 21 ~ 77 days) since no confirmed wound closure occurred after 12 weeks.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TWB-103
Number analyzed (Participants) | 10
days
  Time to Target Ulcer Closure within 12 Weeks | 70 [21 to 77]
  Time to Confirmed Ulcer Closure Up to EOS Visit | 70 [21 to 77]

4. Secondary Outcome: Change of Individual Wound Area for up to 12 Weeks.
Description: The surface area of the ulcer was estimated in the manner as follows. The ulcer along with an ulcer measuring ruler (OPSITETM transparent film) was photographed. An OPSITETM transparent film was placed on the wound and the wound area was traced on the film. The images were processed and analyzed using the ImageJ software package. The ImageJ software read the computed tomographic data and calibrated the images automatically.
Time Frame: Week 1~ Week 12
Population: All Subject Population.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | TWB-103
Number analyzed (Participants) | 10
cm^2
  Baseline | 2.78 (2.124)
  Adjusted Visit 14 (Week 12) with LOCF | 0.52 (0.904)
  Net Change | -2.26 (1.941)

5. Secondary Outcome: Change of Wound Area at Each Week up to 12 Weeks.
Description: as for outcome 4
Time Frame: Week 1 ~ Week 12
Population: All Subject Population.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | TWB-103
Number analyzed (Participants) | 10
cm^2
  Baseline | 2.78 (2.124)
  Adjusted Visit 3 (Week 1) with LOCF | 2.19 (1.963)
  Adjusted Visit 4 (Week 2) with LOCF | 1.65 (1.728)
  Adjusted Visit 5 (Week 3) with LOCF | 1.70 (1.569)
  Adjusted Visit 6 (Week 4) with LOCF | 1.40 (1.531)
  Adjusted Visit 7 (Week 5) with LOCF | 1.21 (1.420)
  Adjusted Visit 8 (Week 6) with LOCF | 1.09 (1.421)
  Adjusted Visit 9 (Week 7) with LOCF | 1.00 (1.380)
  Adjusted Visit 10 (Week 8) with LOCF | 0.75 (1.183)
  Adjusted Visit 11 (Week 9) with LOCF | 0.62 (1.058)
  Adjusted Visit 12 (Week 10) with LOCF | 0.68 (0.944)
  Adjusted Visit 13 (Week 11) with LOCF | 0.96 (1.469)
  Adjusted Visit 14 (Week 12) with LOCF | 0.52 (0.904)

6. Secondary Outcome: General Granulation Rate.
Description: The granulation rate was recorded by comments from the investigator. Healthy granulation tissue was pink to red, moist and shiny. Forming of healthy granulation tissue provided foundation for epithelialization and was an indicator of healing.
Time Frame: Week 1 ~ Week 12
Population: Data were not collected.
Arm/Group | TWB-103
Number analyzed (Participants) | 0

7. Secondary Outcome: Quality of Granulation.
Description: The quality of granulation tissue was recorded by comments from the investigator. Healthy granulation tissue was pink to red, moist and shiny. Forming of healthy granulation tissue provided foundation for epithelialization and was an indicator of healing.
Time Frame: Week 1 ~ Week 12
Population: Data were not collected.
Arm/Group | TWB-103
Number analyzed (Participants) | 0

8. Secondary Outcome: Change of Wound Volume for Individual Subject Measured by 3D Camera and Analysis Software up to 12 Weeks.
Description: For changes of (if data available) wound volume measured by the 3D camera from the baseline values, data was analyzed using one-sample t-test or Wilcoxon sign rank test. (Only for those subjects who have received the 3D measurement)
Time Frame: Week 1 ~ Week 12
Population: There was only one measurement which was performed for one subject at Visit 8.
Measure: Median (Inter-Quartile Range); unit: cm^3
Arm/Group | TWB-103
Number analyzed (Participants) | 1
cm^3 | 0.11 [0.11 to 0.11]

ADVERSE EVENTS:
Time Frame: Day 1 ~ Day 169
Description: The following events were discussed specifically: 1. Study wound and its periphery: Infection, pain, pruritus/irritation, skin dysfunction/blister, osteomyelitis, cellulitis, edema/swelling and unexpected surgery. 2. Non-study area and systemic: Infection, pain, pruritus/irritation, skin dysfunction/blister, osteomyelitis, cellulitis, edema/swelling, unexpected surgery, accidental injury, abnormal lab test and general disorders.
Arm/Group | TWB-103
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TWB-103 (N=10)
Coronary artery disease (Cardiac disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TWB-103 (N=10)
Coronary artery disease (Cardiac disorders) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Application site erosion (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (2)
Anaphylactic shock (Immune system disorders) | 1 (1)
Application site cellulitis (Infections and infestations) | 1 (1)
Application site infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Sweat gland disorder (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT03624023/Prot_SAP_000.pdf